CLINICAL TRIAL: NCT06623578
Title: Comparative Study of Transaxillary Robotic Thyroidectomy With Modified Radical Neck Dissection Versus Conventional Open Surgery in Patients With Papillary Thyroid Carcinoma and Lateral Neck Node Metastases: a Prospective Multicenter Randomized Controlled Study
Brief Title: Comparative Study of Transaxillary Robotic Thyroidectomy With MRND Versus Conventional Open Surgery in N1b PTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2024-495-02
Record Dates: First submitted 2024-09-20; First posted 2024-10-02 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Papillary Thyroid Carcinoma; Lymphatic Metastasis
MeSH Terms: conditions — Thyroid Cancer, Papillary; Lymphatic Metastasis | interventions — Robotic Surgical Procedures; Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robotic-assisted surgery (Experimental)
  Interventions: Procedure: robotic-assisted surgery
- Open Surgery (Other): conventional treatment
  Interventions: Procedure: Open Surgery

INTERVENTIONS:
Procedure: robotic-assisted surgery — robotic-assisted surgery via single-incision transaxillary approach
  Arms: robotic-assisted surgery
Procedure: Open Surgery — conventional open surgery
  Arms: Open Surgery

SUMMARY:
Thyroid cancer is one of the most common malignant tumors in women, ranking seventh in the United States and fourth in China. Papillary thyroid carcinoma is the most common pathological type (about 85% to 90% of thyroid cancers), and lateral cervical lymph node metastasis can reach 0.6-37.5% at diagnosis. For papillary thyroid cancer with lateral cervical lymph node metastasis, the 2015 ATA Guidelines in the United States recommend surgical resection and neck lymph node dissection as the primary treatment. Traditional cervical lymph node dissection often leaves obvious scars in the neck, which seriously affects the postoperative quality of life of patients. The previous studies have shown that endoscopy-assisted surgery with external cervical approach can achieve oncologic effects similar to traditional open surgery in the treatment of N1b papillary thyroid cancer, and can obtain better aesthetic results. However, endoscopic surgery still has some shortcomings, such as poor exposure of some surgical areas and difficult operation. Since November 2016, the investigators tried to apply modified transaxillary robotic-assisted surgery technology to the treatment of thyroid papillary carcinoma in China. The preliminary study included 30 patients, and the results showed that robot-assisted surgery via combined transaxillary-retroaural approach in the treatment of N1b papillary thyroid carcinoma achieved a good oncologic effect (5-year overall survival rate was 100.0%). As the surgical techniques improved, now the investigators can complete robotic-assisted lateral neck lymph node dissection via single-incision transaxillary approach. However, there is still a lack of high-quality evidence on the long-term oncologic outcome and quality of life of this procedure. In this study, a prospective, multi-center, randomized controlled study was conducted to compare the safety, long-term oncologic outcomes and postoperative quality of life of the robot-assisted surgery via single-incision transaxillary approach and open surgery in the treatment of N1b papillary thyroid cancer, which may provide an alternative for the patients with N1b papillary thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old, male or female;
* papillary thyroid carcinoma with ipsilateral lateral cervical lymph node metastasis confirmed by FNAB;
* thyroid tumor of less than 3.0 cm in the largest diameter;
* lack of extrathyroidal extensions as estimated by preoperative ultrasonography and CT.

Exclusion Criteria:

* level I or contralateral neck node metastases.
* enlarged lymph node of larger than 2.0 cm in the short diameter.
* suspected perinodal infiltration of metastatic lymph nodes.
* cervical or/and thoracic deformity.
* life-threatening diseases of liver, kidney, heart and other organs, or abnormal coagulation function.
* clinical evidence of distant metastases such as in the lung, bone, and so on.
* history of previous neck surgery and/or radiation therapy.
* intolerable to general anesthesia
* refuse either surgical procedure
* unwilling to cooperate with long-term follow-up evaluation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
the disease-free survival rate | 60 months
  The 5-year survival rate without a functional, structural, or biological event
Postoperative quality of life：36-Item Short-Form Survey | 12 months
  The quality of life is assessed by 36-Item Short-Form Survey (SF-36) 1 year after surgery, and the differences in physical and physiological dimensions between the two groups were compared. The higher scores mean a better outcome.

SECONDARY OUTCOMES:
Overall survival（OS） | 60 months
  The time from randomization to death from any cause
The dynamic change trend of shoulder function | 60 months
  Shoulder function is assessed using arm abduction test (0-5) to explore the dynamic change. The higher scores mean a better outcome.
The dynamic change trend of the postoperative quality of life | 60 months
  The postoperative quality of life is assessed using 36-Item Short-Form Survey to explore the dynamic change. The higher scores mean a better outcome.
The dynamic change of swallowing function | 60 months
  Swallowing function is assessed using Swallowing Impairment Index 6 (0-24) to explore the dynamic change. The higher scores mean a worse outcome.
The dynamic change trend of neck function | 60 months
  Neck function is assessed using Ten-item Neck Dissection Impairment Index (0-100) to explore the dynamic change. The higher scores mean a better outcome.
The dynamic change trend of aesthetic satisfaction | 60 months
  Aesthetic satisfaction is assessed using verbal response scale (0-10) to explore the dynamic change. The higher scores mean a better outcome.
The dynamic change trend of voice function | 60 months
  Voice function is assessed using Voice Handicap Index 10 (0-40) to explore the dynamic change. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China